CLINICAL TRIAL: NCT00348348
Title: A Study to Evaluate the Clinical and Microbial Efficacy of 0.6% ISV-403 Compared to Vigamox in the Treatment of Bacterial Conjunctivitis
Brief Title: A Study to Investigate the Safety and Efficacy of BOL-303224 in the Treatment of Bacterial Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 434
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Results first posted 2009-08-13 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Acute Bacterial Conjunctivitis
MeSH Terms: interventions — besifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin solution (Active Comparator): Moxifloxacin hydrochloride ophthalmic solution 0.5%
  Interventions: Drug: Moxifloxacin solution
- Besifloxacin Suspension (Experimental): Besifloxacin hydrochloride ophthalmic suspension 0.6%
  Interventions: Drug: Besifloxacin

INTERVENTIONS:
Drug: Besifloxacin — Besifloxacin hydrochloride ophthalmic suspension, 0.6% as base, administered TID for 5 days
  Arms: Besifloxacin Suspension
Drug: Moxifloxacin solution — Moxifloxacin hydrochloride ophthalmic solution 0.5% administered TID for 5 days.
  Arms: Moxifloxacin solution

SUMMARY:
This is a study to investigate a novel drug candidate for the treatment of bacterial conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute bacterial conjunctivitis and exhibit purulent conjunctival discharge and redness in at least one eye.

Exclusion Criteria:

* Pregnant or nursing females.
* Use of any antibiotic within 72 hours of enrollment.
* Any disease conditions that could interfere with the safety and efficacy evaluations of the study drug.
* Participation in an ophthalmic drug or device research study within 30 days prior to entry into this study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1161 (Actual)
Dates: Start 2006-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Comstock, OD, Study Director — Bausch & Lomb Incorporated

REFERENCES:
- [Derived] DeCory HH, Sanfilippo CM, Proskin HM, Blondeau JM. Characterization of baseline polybacterial versus monobacterial infections in three randomized controlled bacterial conjunctivitis trials and microbial outcomes with besifloxacin ophthalmic suspension 0.6. PLoS One. 2020 Aug 25;15(8):e0237603. doi: 10.1371/journal.pone.0237603. eCollection 2020. PMID 32841261
- [Derived] Comstock TL, Paterno MR, Decory HH, Usner DW. Safety and tolerability of besifloxacin ophthalmic suspension 0.6% in the treatment of bacterial conjunctivitis: data from six clinical and phase I safety studies. Clin Drug Investig. 2010;30(10):675-85. doi: 10.2165/11536720-000000000-00000. PMID 20629472

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 84 sites in the US and Asia. First subject was enrolled 6/6/06, and last subject visit was 7/13/07.
Pre-assignment Details: 1161 participants were randomized of which 533 had culture confirmed bacterial conjunctivitis.
Groups:
- Besifloxacin Suspension: Besifloxacin ophthalmic suspension 0.6%
Period: Overall Study
Arm/Group | Moxifloxacin Solution | Besifloxacin Suspension
Started | 579 (Received at least one drop of study medication (Safety Population)) | 582 (Received at least one drop of study medication(Safety Population))
Completed | 554 | 555
Not Completed | 25 | 27
Not completed — Adverse event - unrelated to study drug | 0 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 8 | 10
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Other | 7 | 4
Not completed — Dissallowed Meds - unrelated to study | 1 | 3
Not completed — Dissallowed Meds - unlikley related | 1 | 1
Not completed — Dissallowed Meds - possibly releated | 1 | 1
Not completed — Worsening of BC - Unrelated to study | 0 | 3
Not completed — Worsening of BC - Unlikely related | 1 | 2
Not completed — Adverse event probably related to study | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxifloxacin Solution | Besifloxacin Suspension | Total
Number analyzed (Participants) | 579 | 582 | 1161
Age, Customized [Number; unit: participants]
  <2 years | 15 | 22 | 37
  2 to 9 years | 90 | 91 | 181
  10 to 19 years | 81 | 75 | 156
  20 to 29 years | 73 | 93 | 166
  30 to 39 years | 76 | 71 | 147
  40 to 49 years | 59 | 68 | 127
  50 to 59 years | 65 | 63 | 128
  >/= 60 years | 120 | 99 | 219
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 323 | 332 | 655
  Male | 256 | 250 | 506
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan Native | 6 | 3 | 9
  Asian | 89 | 87 | 176
  Black or African American | 63 | 73 | 136
  Native Hawaiian or Pacific Islander | 2 | 5 | 7
  White | 391 | 385 | 776
  Other | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: Clinical Resolution
Description: Resolution of conjunctival discharge and bulbar conjunctival injection. (mITT, culture confirmed, as treated)
Time Frame: Day 5(+/- 1 day)
Population: modified intent to treat (mITT), culture confirmed, as treated
Measure: Number; unit: Participants
Arm/Group | Moxifloxacin Solution | Besifloxacin Suspension
Number analyzed (Participants) | 281 | 252
Participants | 167 | 147

2. Primary Outcome: Microbial Eradication
Description: eradication of baseline bacterial infection. modified intent to treat (mITT), culture confirmed, as treated
Time Frame: Day 5 (+/- 1 day)
Population: modified intent to treat (mITT), culture confirmed, as treated
Measure: Number; unit: Participants
Arm/Group | Moxifloxacin Solution | Besifloxacin Suspension
Number analyzed (Participants) | 281 | 252
Participants | 256 | 235

3. Secondary Outcome: Clinical Resolution
Description: Clinical resolution of conjunctival discharge and bulbar conjunctival injection, modified intent to treat (mITT), culture confirmed, as treated
Time Frame: Day 8 or Day 9
Population: modified intent to treat (mITT), culture confirmed, as treated
Measure: Number; unit: Participants
Arm/Group | Moxifloxacin Solution | Besifloxacin Suspension
Number analyzed (Participants) | 281 | 252
Participants | 236 | 213

4. Secondary Outcome: Microbial Eradication
Description: Microbial eradication of baseline bacterial infection. modified intent to treat (mITT), culture confirmed, as treated
Time Frame: Day 8 or Day 9
Population: modified intent to treat (mITT), culture confirmed, as treated
Measure: Number; unit: Participants
Arm/Group | Moxifloxacin Solution | Besifloxacin Suspension
Number analyzed (Participants) | 281 | 252
Participants | 238 | 220

ADVERSE EVENTS:
Time Frame: Participants were treated three times daily for 5 days
Description: Safety population - All treated eyes
Arm/Group | Moxifloxacin Solution | Besifloxacin Suspension
Serious Adverse Events (participants affected / at risk) | 1/579 | 1/582
Other Adverse Events (participants affected / at risk) | 0/855 | 0/865
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxifloxacin Solution (N=579) | Besifloxacin Suspension (N=582)
Acute viral syndrome (Infections and infestations) | 1 (1) | 1 (1) — Unlikely related to treatment
Congestive heart failure (Cardiac disorders) | 1 (1) | 1 (1) — Considered unrelated to therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has 45 days to review materials and provide comments back to the investigator.